CLINICAL TRIAL: NCT02338713
Title: A Single-Sequence, 2-Period, Open-Label Study of a Novel Calcium 500 mg and Vitamin D3 1000 IU Chewable Tablet Dosed for 3 Days to Investigate the Effect on Intestinal Calcium Absorption in Healthy Postmenopausal Women and Healthy Men
Brief Title: Effect of Calcium 500 mg and Vitamin D3 1000 IU Chewable Tablet on Intestinal Calcium Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Calcichew-1001; U1111-1163-1751 (Registry Identifier: WHO); 2014-003875-53 (EudraCT Number)
Record Dates: First submitted 2014-12-18; First posted 2015-01-14 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noncarbonated Water + Calcichew D3 (Experimental): Noncarbonated water 200 milliliter (mL), orally, once daily on Days 1, 2 and 3 in period 1 (dummy treatment period) followed by Calcichew D3 500 milligram (mg)/1000 international units (IU) (Calcium 500 mg, chewable tablets and vitamin D3 1000 IU, chewable tablets), orally, once daily on Days 4, 5 and 6 in period 2 (study treatment period) of 6 days treatment period.
  Interventions: Drug: Calcichew D3; Drug: Noncarbonated Water

INTERVENTIONS:
Drug: Calcichew D3 — Calcium 500 mg and vitamin D3 1000 IU chewable tablets
Drug: Noncarbonated Water — Noncarbonated water 200 mL

SUMMARY:
The purpose of this study is to demonstrate that the intestinal absorption of calcium from a novel calcium carbonate-vitamin D3 chewable tablet formulation (calcium 500 milligrams (mg) and vitamin D3 1000 International Units (IU)) increases the amount of calcium excreted in urine and decreases parathyroid hormone (PTH) in serum as compared with Baseline.

DETAILED DESCRIPTION:
The drug being tested in this study was called Calcichew D3. Calcichew D3 was being tested to assess how it is processed by the body in healthy men and postmenopausal women. This study looked at lab results in people who take Calcichew D3.

The study enrolled approximately 27 participants. All participants received the same treatment:

• Calcichew D3 (calcium 500 mg and vitamin D3 1000 IU) chewable tablets All participants were asked to take one tablet each morning of the treatment period.

This single-centre trial was conducted in France. The overall time to participate in this study was up to 44 days. Participants made 2 visits to the clinic, including one 7-day period of confinement to the clinic, and were contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy adult male or female participant.
4. Female participants should be postmenopausal (last menses at least 2 years before signing informed consent and follicle-stimulating hormone (FSH) confirming postmenopausal status).
5. The participant is White.
6. Is aged 45 to 70 years, inclusive, at the time of informed consent and study enrollment.
7. Weighs at least 50 kg and has a body mass index (BMI) from 18 to 30 kilogram per square meter (kg/m^2), inclusive at Screening and Day -1.
8. Is a nonsmoker (having abstained from smoking for at least 6 months).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
4. Has a known hypersensitivity to calcium or vitamin D3 or to any of the excipients of the formulation of the Calcichew D3 chewable tablet.
5. Has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of 5 or more units per day) within 5 years prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine. Ethanol consumption within 72 hours prior to Check-in (Day -1) verified by alcohol breath test (Alcotest).
7. Has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table.
8. Has current or recent (within 6 months) gastrointestinal disorder or gastrointestinal surgery (except appendectomy) that would be expected to influence the absorption of drugs and calcium (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [eg, cholecystectomy]).
9. Has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1.
10. Has a positive test result for hepatitis B surface antigen (HBsAg), antibody to hepatitis C virus (anti-HCV), and human immunodeficiency virus (HIV) antibody at Screening.
11. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 21 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).
12. Has poor peripheral venous access.
13. Has donated or lost 450 millileters (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1.
14. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by both the principal investigator and the Takeda medical monitor.
15. Has abnormal Screening or Day -1 laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than (>)2.0 times the upper limit of normal (ULN).
16. Is a practicing vegetarian or vegan.
17. Has a creatinine clearance according to Modification of Diet in Renal Disease equation of less than (<)60 mL/min at Screening or Check-in (Day -1).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Rennes, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in France from 16 January 2015 to 24 February 2015.
Pre-assignment Details: Healthy participants were enrolled in this study. Treatment period of study comprised of 2-periods. Participants received noncarbonated water in period 1 (dummy treatment period) and Calcichew D3 in period 2 (study treatment period).
Groups:
- Noncarbonated Water+Calcichew D3: Noncarbonated water 200 milliliter (mL), orally, once daily on Days 1, 2 and 3 in period 1 (dummy treatment period) followed by Calcichew D3 500 milligram (mg)/1000 international units (IU) (Calcium 500 mg, chewable tablets and vitamin D3 1000 IU, chewable tablets), orally, once daily on Days 4, 5 and 6 in period 2 (study treatment period) of 6 days treatment period.
Period: Overall Study
Arm/Group | Noncarbonated Water+Calcichew D3
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of dummy treatment.
Arm/Group | Noncarbonated Water+Calcichew D3
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.3 (9.16)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 68.0 (11.088)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.49 (2.594)
Smoking classification [Number; unit: participants]
  Never Smoked | 18
  Current Smoker | 0
  Ex-Smoker | 9
Alcohol classification [Number; unit: participants]
  Never Drunk | 22
  Current Drinker (less than 5 units per day) | 5
Xanthine/Caffeine Consumption [Number; unit: participants]
  Had Consumption | 21
  Had no Consumption | 6
Number of Participants who were Postmenopausal [Number; unit: participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: PTH AUC(0-6): Area Under the Serum Concentration-Time Curve From Time 0 to 6 Hours for Parathyroid Hormone
Description: The PTH AUC(0-6) is a measure of the area under the serum concentration-time curve from 0 to 6 hours of parathyroid hormone.
Time Frame: Days 3 and 6: pre-dose and at multiple time-points (upto 6 hours) postdose. Day 3 for the noncarbonated water reporting group and Day 6 for the Calcichew D3 reporting group
Population: The Pharmacodynamic(PD) serum analysis set included all participants who received at least 1 dose of dummy treatment and had at least 1 measurable serum concentration of parathyroid hormone in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram per milliliter (hr*pg/mL)
Groups:
- Noncarbonated Water: Noncarbonated water 200 mL, orally, once daily on Days 1, 2 and 3 in period 1 (dummy treatment period).
- Calcichew D3: Calcichew D3 500 mg/1000 IU (Calcium 500 mg, chewable tablets and vitamin D3 1000 IU, chewable tablets), orally, once daily on Days 4, 5 and 6 in period 2 (study treatment period).
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
hour*picogram per milliliter (hr*pg/mL) | 215 (30.3) | 157 (31.5)

2. Primary Outcome: (Ca^2+ Ae6): Amount of Calcium Excreted in Urine From Time 0 to 6 Hours Post-dose
Description: Ca^2+ Ae6 was calculated as the urine volume of the urine collected from 0 to 6 hours multiplied by the calcium concentration measured in urine.
Time Frame: as for outcome 1
Population: The pharmacokinetic(PK) urine analysis set included all participants who received at least 1 dose of dummy treatment and had at least 1 measurable urine concentration of calcium in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles (mmol)
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
millimoles (mmol) | NA (NA) — No data was reported since Geometric mean was not calculated when minimum value was '0', as predefined in protocol. | 1.74 (40.6)

3. Secondary Outcome: PTH AUC (0-24): Area Under the Serum Concentration-Time Curve From Time 0 to 24 Hours for Parathyroid Hormone
Description: The PTH AUC(0-24) is a measure of the area under the serum concentration-time curve from 0 to 24 hours of parathyroid hormone.
Time Frame: Days 3 and 6: pre-dose and at multiple time-points (up to 24 hours) postdose. Day 3 for the noncarbonated water reporting group and Day 6 for the calcichew D3 reporting group
Population: The PD serum analysis set included all participants who received at least 1 dose of dummy treatment and had at least 1 measurable serum concentration of parathyroid hormone in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
hr*pg/mL | 1020 (30.5) | 908 (29.5)

4. Secondary Outcome: (Ca^2+ Ae24): Amount of Calcium Excreted in Urine From Time 0 to 24 Hours Post-dose
Description: Ca2+ Ae0-24 was calculated as the urine volume of the urine collected from 0 to 24 hours multiplied by the calcium concentration measured in urine.
Time Frame: Days 3 and 6: pre-dose and at multiple time-points (upto 24 hours) postdose. Day 3 for the noncarbonated water reporting group and Day 6 for the Calcichew D3 reporting group
Population: The PK urine analysis set included all participants who received at least 1 dose of dummy treatment and had at least 1 measurable urine concentration of calcium in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
mmol | 3.21 (52.2) | 4.67 (34.6)

5. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for Calcium
Time Frame: Days 3 and 6: predose and at multiple time-points (up to 24 hours) postdose. Day 3 for the non carbonated water reporting group and Day 6 for the Calcichew D3 reporting group
Population: The PK serum analysis set included all participants who received at least 1 dose of dummy treatment and had at least 1 measurable serum concentration of calcium in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles per litre(mmol/L)
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
millimoles per litre(mmol/L) | 2.35 (2.1) | 2.40 (2.9)

6. Secondary Outcome: AUC(0-6): Area Under the Serum Concentration-Time Curve From Time 0 to 6 Hours for Calcium
Time Frame: Days 3 and 6: predose and at multiple time-points (up to 6 hours) postdose. Day 3 for the non carbonated water reporting group and Day 6 for the Calcichew D3 reporting group
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*millimoles per litre (hr*mmol/L)
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
hour*millimoles per litre (hr*mmol/L) | 13.5 (2.3) | 13.9 (2.6)

7. Secondary Outcome: AUC(0-24): Area Under the Serum Concentration-Time Curve From Time 0 to 24 Hours Post-dose for Calcium
Time Frame: as for outcome 5
Population: The PK serum analysis set of included participants who received at least 1 dose of dummy treatment and had at least 1 measurable serum concentration of calcium in each treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*mmol/L
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
hr*mmol/L | 53.8 (2.2) | 55.0 (3.0)

8. Secondary Outcome: Tmax: Time to Reach the Cmax for Calcium
Time Frame: as for outcome 5
Population: The PK analysis set consisted of all participants who received at least 1 dose of dummy treatment and who had at least 1 measurable serum concentration of calcium in each treatment period.
Measure: Median (Full Range); unit: hours
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
hours | 24.0 (8.72) [3.00 to 24.0] | 4.00 (7.45) [0.517 to 24.0]

9. Secondary Outcome: Number of Participants Who Experience at Least 1 Treatment-Emergent Adverse Event (TEAE)
Time Frame: Baseline up to 14 days after last dose of study drug (Day 21)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of dummy treatment.
Measure: Number; unit: participants
Arm/Group | Noncarbonated Water | Calcichew D3
Number analyzed (Participants) | 27 | 27
participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 14 days after the last dose of Calcichew D3 study drug (21 days).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Noncarbonated Water | Calcichew D3
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noncarbonated Water (N=27) | Calcichew D3 (N=27)
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.